CLINICAL TRIAL: NCT06639269
Title: Effect of Fertility Health Education Program Given to Young People on Fertility Health Knowledge and Healthy Life Awareness: Randomized Controlled Study
Brief Title: Effect of Fertility Health Education Program on Fertility Health Knowledge and Healthy Life Awareness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Rabia ERKAN KIRMIZIGÜL, REGISTERED NURSE, PhD student, Ankara University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AU-IHS-REK-01
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Youth; Education; Fertility
Keywords: youth; education; Fertility Health Information; Healthy Life Awareness
MeSH Terms: interventions — Early Intervention, Educational

STUDY DESIGN:
Intervention Model Description: In our study, we will have two groups: control and intervention. A 3-session fertility health education program will be applied to the students in the intervention group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): All those who remain will be asked to fill out the Introductory Information Form, Fertility Health Information Scale and Healthy Life Awareness Scale during the pre-test phase.
  6 weeks after the pre-test, the authorized person in the control groups will be contacted and expected to complete the Fertility Health Information Scale and Healthy Life Awareness Scale.
  The control group will not receive training.
- educational program intervention group (Experimental): The "Fertility Health Education Program", which will be created in line with literature information, will be applied to the intervention group. Participants selected for the intervention group will be divided into groups of 10-15 people. Participants in each group will be informed about the date, time and location of the education program through methods suitable for the student; e-mail, phone or message. The education program will consist of 3 sessions. Education sessions will be planned on days and times when the researcher, classrooms and students are available. For students who cannot attend group education, make-up education will be provided within a week. In this study, the interval between sessions will be planned as 1 week. Group education will be planned according to the times when the students are available. PowerPoint presentation, models, booklets and brochures will be used in the education sessions.
  Interventions: Other: fertility health education program

INTERVENTIONS:
Other: fertility health education program — The intervention group will be implemented with a "fertility health education program" for which a literature information document will be created. In the training; booklets and brochures will be prepared. The control unit will include information on programming and data collection forms to be used. Those selected from the intervention group will be divided into groups of 10-15 people. The training program will consist of 3 sessions. Training sessions will be planned on days and hours that are convenient for the researcher, classrooms and students. For students who cannot attend group training, make-up training will be provided within a week. In this study, the time between sessions will be planned as 1 week. The sessions in this study will be planned to be in groups of 10-15 people and will last 50 minutes.
  Other Names: fertility health education; education program
  Arms: educational program intervention group

SUMMARY:
This study was planned to examine the effect of the fertility health education program given to young people on fertility health knowledge and healthy life awareness.

The study was planned to be conducted as a randomized controlled experimental study in the pre-test-post-test order.

The population of the research will consist of students studying at Gaziantep University Naci Topçuoğlu Vocational School in the 2024-2025 academic year. The research sample was calculated as a minimum of 64 people per group (experimental and control group) and 128 people in total. Considering the possible losses that may occur during the research process, a total of 146 students are planned to be accepted.

Data in the research; It will be collected through "Introductory Information Form", "Fertility Health Information Scale", "Healthy Life Awareness Scale" and "Training Program Satisfaction Survey".

In the research, the Fertility Health Education Program consisting of 3 sessions will be applied to the intervention group, and the control group will be informed about the research process and the data collection forms to be used. Data collection forms will be applied to students in both groups before and after the training.

In the analysis of the data; mean±standard deviation and median (minimum-maximum) will be used for quantitative variables as descriptors, and the number of patients (percentage) will be used for qualitative variables.

Student-t test, Mann-Whitney U test, One Way ANOVA test, Kruskal Wallis H test, Chi-square and Fisher exact tests will be used in the analysis, depending on the assumption of normal distribution. Risk factors affecting the qualitative dependent variable will be examined with Logistic Regression analysis. The statistical significance level will be taken as 0.05.

DETAILED DESCRIPTION:
The study is planned to be conducted in three stages: first stage (pre-intervention), second stage (intervention) and third stage (post-intervention). First Stage (Pre-Intervention): Students studying at the Vocational School where the study will be conducted will be informed about the study and invited to participate in the study. A list of students who meet the inclusion criteria and agree to participate in the study will be created. The gender and phone numbers of the students will be recorded while creating the list. The list will be sent to a statistician to determine the intervention and control groups using the randomization method. Students will be randomized into the intervention and control groups with similar gender distribution. Consent will be obtained from the participants included in the study through the Informed Consent Form.

Second Stage (Intervention): The "Fertility Health Education Program", which will be developed in line with literature information, will be applied to the intervention group. Both the pre-test and the first session of the training will be held on the same day. All participants will be asked to fill out the Introductory Information Form, Fertility Health Information Scale and Healthy Life Awareness Scale during the pre-test stage.

Third Phase (Post-Intervention): In this study, the post-test is planned to be administered 4 weeks after the last training. In order to complete the post-test, students in the intervention group will be contacted 4 weeks after the last training and the control group will be contacted 6 weeks after the pre-test and the Fertility Health Knowledge Scale and Healthy Life Awareness Scale will be completed.

In order to conduct the research, permission was obtained from Ankara University Ethics Committee with the decision numbered 06/04 and dated 03.04.2024, and in order to collect the research data, permission was obtained from Gaziantep University Naci Topçuoğlu Vocational School, where the research will be conducted, dated 02.09.2024 and numbered E-87841438-100-539736. Data collection forms will be distributed to the volunteers by the researcher, and the forms will be filled in by the volunteers. While filling out the forms, a distanced seating arrangement will be created so that the volunteers cannot see each other's answers. The data obtained from the research will be analyzed anonymously and the confidentiality of the data will be ensured. The research will be conducted in accordance with the Declaration of Helsinki. The researcher will inform the students who make up the sample that participation in the research is voluntary and that they can withdraw from the research at any time, and the purpose and method of the research will be explained. In addition to their verbal consent, students who agree to participate in the research will be asked to sign an Informed Consent Form. After the completion of the research, students in the control group who want to receive training and students who volunteer to participate in the study but cannot be in the intervention or control groups and want to receive training will be given a single session of fertility health training, an education booklet will be distributed, and a brochure will be sent to their phones.

ELIGIBILITY:
Inclusion Criteria:

1. Between the ages of 18-24,
2. Unmarried,
3. Not having children,
4. Not being pregnant or having a pregnant partner (for men)
5. Not having a condition that would prevent communication (visual, hearing impairment, etc.),
6. Not working on education regarding fertility health and/or healthy living awareness,
7. Not having chronic children,
8. Volunteers to participate in the research.

Exclusion Criteria:

1. Those who could not continue the research for any reason,
2. Those who did not participate in all the implemented initiatives,
3. Those who did not fill out the data collection tools.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 133 (Actual)
Dates: Start 2024-10-14 (Actual); Primary Completion 2024-12-13 (Actual); Study Completion 2024-12-14 (Actual)

PRIMARY OUTCOMES:
Fertility Health Information Level | 6 months
  Fertility Health Information Scale. The scale consists of 30 items and has a single factor structure. Responses to the items related to the scale are in the five-point Likert type (5-definitely yes; 4-probably yes; 3-undecided; 2-probably no; 1-definitely no). The 20th item is reverse coded in the evaluation. Then, the responses are classified as "correct" or "incorrect". Those who mark the option "definitely yes" and "probably yes" are accepted as correct. The knowledge level is expressed as a percentage based on the scale items and their total.
Healthy Life Awareness | 6 months
  Healthy Life Awareness Scale is a 5-point Likert-type scale consisting of 4 sub-dimensions and 15 items. It consists of the sub-dimensions of change (items 1-5), socialization (items 6-9), responsibility (items 10-12), and nutrition (items 13-15). The lowest score to be obtained from the scale is 15, the highest score is 75. A high score from the scale is evaluated as a high level of healthy life awareness.

CONTACTS AND LOCATIONS:
Overall Officials: Funda Ozdemir, Assoc. Prof., Study Director — Ankara University
Locations (1):
- Gaziantep University, Naci Topçuoğlu Vocational School, Gaziantep, Şehitkamil, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No